CLINICAL TRIAL: NCT06380621
Title: A Comparative Longitudinal Study Between Bilateral Totally Extraperitoneal Repair and Unilateral Totally Extraperitoneal Repair Among Patients of Unilateral Inguinal Hernia at a Tertiary Care Hospital in Eastern Nepal
Brief Title: Bilateral vs Unilateral Totally Extraperitoneal Repair Among Patients With Unilateral Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Bikash kumar sah, Lecture (General Surgery), B.P. Koirala Institute of Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRC/1386/018
Record Dates: First submitted 2024-03-16; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Inguinal Hernia
Keywords: totally extra peritoneal (TEP)repair; Occult contralateral hernia; Inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — tetraethylpyrazine; Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bilateral TEP group (Experimental): Bilateral TEP repair
  Interventions: Procedure: Totally Extra Peritoneal repair (TEP) repair
- Unilateral TEP group (Active Comparator): Unilateral TEP repair
  Interventions: Procedure: Totally Extra Peritoneal repair (TEP) repair

INTERVENTIONS:
Procedure: Totally Extra Peritoneal repair (TEP) repair — TEP repair

SUMMARY:
The goal of this clinical trial is to investigate the feasibility of bilateral laparoscopic exploration for all unilateral cases followed by laparoscopic bilateral TEP repair in all cases with a contralateral occult hernia and to compare complications, recurrence rates, postoperative pain, and operative duration with prospectively performed unilateral repairs in young to middle-aged patients presenting with unilateral hernias in the surgery outpatient department.

The main questions it aims to answer are:

* To compare complications, recurrence rates, postoperative pain, and operative duration between both groups.
* Incidence of occult contralateral hernia Patients attending the OPD for unilateral inguinal hernia were counseled about the trial and fully encouraged to understand the difference between two procedures for unilateral hernia: bilateral exploration and bilateral TEP repair, upon which if a contralateral occult inguinal hernia was observed, documented, and controls were taken from the patients who denied bilateral exploration and underwent unilateral TEP repair. The allotment of patients was done in two groups of 30 patients each.

Researchers will compare Group A( bilateral TEP) with Group B (unilateral TEP) to see if complications, recurrence rates, postoperative pain, and operative duration occur in each group

DETAILED DESCRIPTION:
Introduction Today, laparoscopic total extraperitoneal (TEP) surgery has emerged as the preferred and standard approach in today's era of technology, owing to the various benefits of laparoscopic surgery. Patients with unilateral inguinal hernia have a lifetime risk of 33% of developing hernia on the contralateral side.1 A study by Bochkarev, V. and Lal, P. et al. showed approximately 22% of bilateral defects in patients with unilateral inguinal hernia at TEP. 2,3 Another study found reasonable (20-25%) chance of discovering an occult contralateral hernia on exploration of the clinically asymptomatic side in unilateral hernias.3 Moreover, Studies have reported an incidence rate of 5%-58% for occult contralateral hernias at the time.4 The patient is at high risk of fibrous adhesions, bowel and bladder injury, and port site hernia if repeat TEP is planned for contralateral inguinal hernia repair. Thus, performing a bilateral repair for a unilateral hernia with/without an occult contralateral defect renders the patient free of the possibility of developing a contralateral primary inguinal hernia later in life, and this can be done in a single sitting or a single hospital stay. The patient holds various benefits (decreased chances of repeat anesthesia-related complications, risk of intra-peritoneal adhesions, bowel perforation, monitoring advantage) except for a minor increase in surgery time.5

Laparoscopic inguinal hernia repair is the standard procedure in our department and is highly demanding, complex, and at times controversial. No data is available till date regarding operative duration, complications, and recurrence rates in the Nepalese population. So, this study is designed to evaluate the constraints of this problem in the context of our developing country, measuring the outcomes between these two groups. The purpose of this study is to have a specific management plan for laparoscopic inguinal hernia repair, provide rationale for a current management plan, and try to formulate a protocol for our hospital. Whether clinically diagnosed unilateral inguinal hernias allow bilateral exploration, a bilateral repair would benefit the patient in the long term or not, and we anticipate evolving policy changes in the days ahead.

Method:

A total of 60 patients were included in this prospective longitudinal study from March 2018 to March 2019. Patients attending the OPD for unilateral inguinal hernia were counseled about the trial. Patients who gave consent for bilateral inguinal exploration and repair were kept in Group A, and those who did not consent for bilateral exploration and underwent unilateral repair were kept in Group B. The allotment of patients was done in two groups of 30 patients each.

ELIGIBILITY:
Inclusion Criteria:

1. age group of 16-55 years
2. clinically diagnosed unilateral inguinal hernia

Exclusion Criteria:

1. complicated hernia (obstructed and strangulated);
2. past history of pelvic radiotherapy
3. patient unfit for general anesthesia; and
4. patient not giving consent

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
To compare pain in between patients of bilateral totally extra peritoneal repair and unilateral totally extra peritoneal repair. | 6 months
  The postoperative pain was recorded by a pictorial Visual Analogue Scale (VAS) at 6 hours, 12 hours, and 24 hours during the hospital stay, and during follow up in the outpatient department on the 10th day, 1 month, 3 months, and 6 months, respectively.
To measure incidence of intra- and post-operative complication between patients of unilateral and bilateral TEP repair | 6 months
  intraoperative complications: Visceral injury, Subcutaneous emphysema Postoperative: seroma, wound infection, and recurrence assessed during the hospital stay and during follow-up in the outpatient department on the 10th day, 1 month, 3 months, and 6 months, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh kumar Gupta, Ms, Principal Investigator — B. P. Koirala institute of health science
Locations (1):
- Bikash Kumar Sah, Dharān, Koshi, Nepal

REFERENCES:
- [Background] Kara H, Arikan AE, Dulgeroglu O, Moldur DE, Uras C. Management of Occult Contralateral Inguinal Hernia: Diagnosis and Treatment With Laparoscopic Totally Extra Peritoneal Repair. Surg Laparosc Endosc Percutan Tech. 2020 Jun;30(3):245-248. doi: 10.1097/SLE.0000000000000765. PMID 32032331
- [Background] Bochkarev V, Ringley C, Vitamvas M, Oleynikov D. Bilateral laparoscopic inguinal hernia repair in patients with occult contralateral inguinal defects. Surg Endosc. 2007 May;21(5):734-6. doi: 10.1007/s00464-007-9196-x. Epub 2007 Feb 20. PMID 17310298
- [Background] Pawanindra Lal, Philips P, Chander J, Ramteke VK. Is unilateral laparoscopic TEP inguinal hernia repair a job half done? The case for bilateral repair. Surg Endosc. 2010 Jul;24(7):1737-45. doi: 10.1007/s00464-009-0841-4. Epub 2010 Feb 5. PMID 20135181
- [Background] Tiwary SK, Kumar S, More R, Shankar V, Kumar S, Dwivedi AND. A study of contralateral occult inguinal hernia in adult male patients undergoing total extraperitoneal herniorraphy. J Family Med Prim Care. 2020 Jun 30;9(6):2975-2979. doi: 10.4103/jfmpc.jfmpc_207_20. eCollection 2020 Jun. PMID 32984158
- [Background] Kockerling F, Schug-Pass C, Adolf D, Keller T, Kuthe A. Bilateral and Unilateral Total Extraperitoneal Inguinal Hernia Repair (TEP) have Equivalent Early Outcomes: Analysis of 9395 Cases. World J Surg. 2015 Aug;39(8):1887-94. doi: 10.1007/s00268-015-3055-z. PMID 25832474

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT06380621/Prot_ICF_000.pdf